CLINICAL TRIAL: NCT02403141
Title: Abu Dhabi Sleep Apnea (ADSA) Study
Acronym: ADSA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Imperial College London Diabetes Centre (Other)
Responsible Party: Principal Investigator, Dr Nader Lessan, MD, Consultant Endocrinologist, Imperial College London Diabetes Centre
Other Study IDs: IREC020
Record Dates: First submitted 2015-03-25; First posted 2015-03-31 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Sleep Apnoea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Normal glucose tolerance: Patients with normal fasting glucose. Blood glucose less than 5.6mmol/L
  Interventions: Other: Questionnaire
- Impaired fasting glycaemia: Patients with blood glucose between 5.6mmol/L - 7mmol/L
  Interventions: Other: Questionnaire
- Type 2 diabetes: Patients with blood glucose higher than 7mmol/L and negative IA2 and GAD antibodies.
  Interventions: Other: Questionnaire
- Type 1 diabetes: Patients on insulin and with positive IA2 and/or GAD antibodies.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire

SUMMARY:
Obstructive sleep apnoea (OSA) is a common medical problem which, despite increasing awareness, remains under-diagnosed. There is a close association between OSA and obesity; 60-70% of patients diagnosed with OSA are either obese or overweight [1]. OSA is also very common among patients with type 2 diabetes. Type 2 Diabetes Mellitus (T2DM) has reached epidemic status in the Gulf region. OSA worsens insulin resistance and leads to weight gain through sleep disturbance [2]. Several mechanisms have been proposed for the associations of OSA with diabetes and obesity [3]. At present there is little available information regarding the prevalence of OSA in the UAE, the relationship with T2DM and obesity, and the impact of OSA on health outcomes in the Emirati population. This research will explore these relationships and inform public health decisions regarding diagnostic pathways, service provision and treatment protocols.

ELIGIBILITY:
Inclusion Criteria:

Participants aged between 18-64 years old. Both Gender male and female.

Exclusion Criteria:

Paediatrics below the age of 18. Any participant who is unable to take part

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients over the age of 18 attending ICLDC will be offered the option of taking part in the study. Those agreeing to participate will be asked to fill in a questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Primary objective (Establishing the prevalence of OSA in the study population.) | 3 months
  Establishing the prevalence of OSA in the study population.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London Diabetes Centre, Abu Dhabi, United Arab Emirates